CLINICAL TRIAL: NCT03789682
Title: Predictive Value of CD155 for Survival and Effectiveness of Chemotherapy in Patients With Muscle Invasive Bladder Cancer
Brief Title: CD155 in Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bo Dai, Department of Urology, Fudan University
Other Study IDs: FUSCC-URO1201-2018-1
Record Dates: First submitted 2018-12-27; First posted 2018-12-28 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FUSCC cystectomy cohort: patients underwent cystectomy in Fudan University Shanghai Cancer Center
  Interventions: Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Adjuvant chemotherapy — adjuvant chemotherapy using Gemcitabine plus Cisplatin

SUMMARY:
This research is designed to investigate the prognostic and predictive value of CD155 in muscle invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-metastatic muscle invasive bladder cancer
* pathology confirmed urothelial carcinoma
* underwent cystectomy and pelvic lymph node dissection

Exclusion Criteria:

* not enough tissue for immunohistochemistry
* patients with a second neoplasm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-metastatic muscle invasive bladder cancer underwent cystectomy in Fudan University Shanghai Cancer Center is included
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Recurrence free survival | 2018.1.1-2023.12.31
  Time to recurrence or metastasis

SECONDARY OUTCOMES:
Overall survival | 2018.1.1-2028.1.1
  Time to death
Benefit from neoadjuvant chemotherapy | 2018.1.1-2028.1.1
  response to neoadjuvant chemotherapy
Benefit from adjuvant chemotherapy | 2018.1.1-2028.1.1
  Survival analysis grouped by adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided